CLINICAL TRIAL: NCT04553874
Title: Health Status of the Oldest-old Population: a Population-based, Cohort Study
Brief Title: Health Status of the Oldest-old Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Chun Zhang, professor, Peking University
Other Study IDs: IRB00006761-M2020021
Record Dates: First submitted 2020-09-12; First posted 2020-09-18 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: the Health Status of the Oldest Old
Keywords: oldest-old; epidemiology; population-based; cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the blood, urine, and stool specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — observational study without intervention

SUMMARY:
This study aims to investigate the health status of the oldest-old population and to explore the key factors associated with their quality of life The study will select all the elderly aged 85 years and above from Lanqiying Community, Qinghuayuan Street, Haidian District, Beijing, and enroll them after informed consent. Demographic, sociological, economic, physiological information and disease-related records will be collected through questionnaire interviews, scales, and examinations.

After the first survey, the participants will be followed for 2 years to collect information about deaths or major health events. The baseline survey will be re-conducted two years later.

DETAILED DESCRIPTION:
This study is a population-based cohort study. Oldest-old people (aged 80 and over) will be enrolled.

Data collection Social economics information include: name, gender, age, nationality, marital status, personal habits, occupation, level of education, family living situation, monthly income, way to go to a doctor and medical payment, etc The health status and disease will be obtained by review the medical records as well as the narration of the subjects and their family members. We will focus on diseases with high disability mortality, high social burden. Multiple indicators or abilities will be evaluated through the scale, including life or acting ability, nutritional status, cognitive ability, psychological status, social support, quality of life self-assessment, etc., so as to comprehensively understand the comprehensive information of the participants.

Basic physical examination and special clinical examination will be performed to obtain multiple objective indicators reflecting the subject's physical function The basic health examination includes; Blood pressure, respiration, heart rate, pulse; Height, weight, waist circumference, hip circumference, arm circumference, calf circumference, grip strength, vital capacity, tooth condition, hearing condition, visual acuity, ECG, etc.

Special examinations include the blood, urine, and stool specimens. Imageological examination like MRI, fundus photography, and optical coherence tomography will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* All the people aged 80 years and above in the target community in Beijing

Exclusion Criteria:

* People who were hospitalized for long period (6 months or more) or at the end of their lives were excluded.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All the people aged 80 years and above in the target community in Beijing will be enrolled, and people who were hospitalized for long period (6 months or more) or at the end of their lives were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Death | 3 years
  The incidence of death during the study period

CONTACTS AND LOCATIONS:
Overall Officials: chun Zhang, doctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hosipital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No